CLINICAL TRIAL: NCT03470480
Title: The Use of Repetitive Transmagnetic Stimulation to Target Craving in Methamphetamine Use Disorder
Brief Title: rTMS for Craving in Methamphetamine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brandon Cornejo MD, PhD, Assistant Professor, Psychiatry, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GPSYC0236A
Record Dates: First submitted 2018-02-07; First posted 2018-03-20 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Methamphetamine Abuse; Substance Use Disorders; Stimulant Dependence; Methamphetamine-dependence; Stimulant Use; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This preliminary study aims to consent and enroll 20 individuals with Methamphetamine Use Disorder. Participants will be randomized into two rTMS conditions (real versus sham) and two picture cues conditions (METH versus neutral). Randomization provides the following four groups: real METH (RM), real neutral (RN), sham METH (SM) and sham neutral (SN). The randomizations can be performed with a web-based randomization generator (www.randomization.com) (47). Subjects and rTMS administrators will be blinded to the treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Treatment rTMS + meth pictures (Experimental): Participants in this group will receive real repetitive transcranial magnetic stimulation treatments. Before each rTMS session they will be exposed to a series of methamphetamine-related pictures to evaluate response to methamphetamine visual cues while receiving real rTMS treatments. This group will be referred to as real METH (RM).
  Interventions: Device: Real Repetitive transcranial magnetic stimulation; Behavioral: Methamphetamine visual cues
- Treatment rTMS + neutral pictures (Active Comparator): Participants in this group will receive real repetitive transcranial magnetic stimulation treatments. Before each rTMS session they will be exposed to a series of neutral pictures to evaluate response to neutral visual cues while receiving real rTMS treatments. This group will be referred to as real neutral (RN).
  Interventions: Device: Real Repetitive transcranial magnetic stimulation; Behavioral: Neutral visual cues
- Sham rTMS + meth pictures (Sham Comparator): Participants in this group will receive sham repetitive transcranial magnetic stimulation treatments. Before each rTMS session they will be exposed to a series of methamphetamine-related pictures to evaluate response to methamphetamine visual cues while receiving sham rTMS treatments. This group will be referred to as sham METH (SM).
  Interventions: Device: Sham Repetitive transcranial magnetic stimulation; Behavioral: Methamphetamine visual cues
- Sham rTMS + neutral pictures (Sham Comparator): Participants in this group will receive sham repetitive transcranial magnetic stimulation treatments. Before each rTMS session they will be exposed to a series of neutral pictures to evaluate response to neutral visual cues while receiving sham rTMS treatments. This group will be referred to as sham neutral (SN).
  Interventions: Device: Sham Repetitive transcranial magnetic stimulation; Behavioral: Neutral visual cues

INTERVENTIONS:
Device: Real Repetitive transcranial magnetic stimulation — A real magnet will be used during rTMS treatments, which will look identical to the sham magnet. The participants and treatment facilitator will be blinded to which magnet will be used. High frequency repetitive transmagnetic stimulation (rTMS) will be directed at left dorsolateral prefrontal cortex (DLPFC) during 10 daily treatments within two weeks then 6 more treatments during the following month.
  Other Names: rTMS; TMS; Magstim Rapid 2
  Arms: Treatment rTMS + meth pictures; Treatment rTMS + neutral pictures
Device: Sham Repetitive transcranial magnetic stimulation — A sham magnet will be used during rTMS treatments, which will look identical to the real magnet. The participants and treatment facilitator will be blinded to which magnet will be used. The sham rTMS treatments will be directed at left dorsolateral prefrontal cortex (DLPFC) during 10 daily treatments within two weeks then 6 more treatments during the following month.
  Arms: Sham rTMS + meth pictures; Sham rTMS + neutral pictures
Behavioral: Methamphetamine visual cues — Just before each rTMS session, participants will be shown methamphetamine-related pictures
  Arms: Sham rTMS + meth pictures; Treatment rTMS + meth pictures
Behavioral: Neutral visual cues — Just before each rTMS session, participants will be shown neutral pictures
  Arms: Sham rTMS + neutral pictures; Treatment rTMS + neutral pictures

SUMMARY:
The primary aim of this project is to use a randomized single-blind sham-controlled study to investigate if high frequency repetitive transmagnetic stimulation (HF-rTMS) can modulate cue-induced craving in adult methamphetamine (METH) users. The investigators hypothesize that HF-rTMS directed at left dorsolateral prefrontal cortex (DLPFC) will result in a reduction in craving for METH compared to sham-controlled rTMS in adults with methamphetamine use disorder (MUD) as evidenced by validated measures of METH craving. Neurobiologically, the investigators anticipate rTMS mediated stimulation of the DLPFC could result in inhibition of cue-induced craving through potential disruption of involved circuitry. The current project proposes that participants who are recently abstinent from METH will be randomized into four experimental groups to provide two rTMS conditions (real versus sham) and two picture cues conditions (METH versus neutral). The experiment will have an induction phase where each subject will receive 10 daily treatments within 2 weeks. Just before each rTMS/sham session participants will be shown visual cues (METH or neutral). Participants will then undergo a maintenance phase for an additional month with assessments to evaluate craving and relapse. Urine samples for urine drug screening (UDS) will be collected at screening day and on days 1, 5 and 10. Just before each rTMS/sham session participants will be shown visual cues (METH and neutral). VAS craving scores will be assessed before and after picture presentation and after the rTMS/sham session. Before the first and 10th treatment session, participants were evaluated by the the Stimulant Craving Questionnaire (STCQ) and the Severity of Dependence Scale (SDS) questionnaires. Participants will then undergo a maintenance phase for an additional month. During the first week of maintenance, three rTMS/sham sessions will be administered. During each of the following 3 weeks, one rTMS/sham session will be given per week. As with the induction phase, urine samples will be collected for screening and STCQ and the SDS questionnaires will be completed at each maintenance session. To evaluate the long-term effects of the rTMS treatment, the investigators plan on contacting participants 6 months after treatment termination for all subjects who completed the 10 treatment sessions. During that phone conversation, craving and relapse will again be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must use at least 0.5 g per day at least 5 days per week and have a minimum 12-month history of METH abuse.
* Subjects must meet DSM V diagnosis for methamphetamine use disorder.
* Subjects must have a minimum 4-week period of detoxification and a desire to stop using methamphetamine.

Exclusion Criteria:

* Present or past history of neurological disorder
* The present history of a DSM IV Axis I or DSM V primary psychiatric disease (apart from MUD and depressive symptoms defined as a Hamilton Depression Scale Score < 7 ("normal"))
* Scores on the Hamilton Depression Scale > 8, possibly indicating clinical depression
* No current abuse of drugs other than methamphetamine (except nicotine). Urine-screening tests for psychoactive drugs will be performed to corroborate the lack of drug use.
* Individuals meeting criteria for cannabis use disorder or alcohol use disorder
* Medical illness that can affect brain function
* Past or present history of cardiovascular disease or high blood pressure
* Any history of epilepsy or a known history of seizure disorder
* A history of metal in the head or chest area (except dental fillings or braces)
* Current consumption of psychiatric medication
* Any other medical, neurological or neurosurgical condition that would preclude the administration of repetitive transmagnetic stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Effect of rTMS directed at left DLPFC on craving for methamphetamine as assessed by the Severity of Dependence Scale. | 6 weeks
  The Severity of Dependence Scale (SDS) is a 5-item questionnaire that provides a score indicating the severity of dependence on methamphetamine. Each of the five items is scored on a 4-point scale (0-3). The total score is obtained through the addition of the 5-item ratings and will range from 0 to 15. The higher the score the higher the level of dependence. Pre and post differences in craving will be assessed.
Effect of rTMS directed at left DLPFC on craving for methamphetamine as assessed by a Visual Analog Scale (VAS). | 6 weeks
  The visual analogue scale (VAS) is a fixed-length horizontal line on which the participant draws a line between the two anchors of "no cravings at all" and "most intense craving imaginable". The distance between the "no cravings at all" anchor and the participants line is measured and reported as a value between 0 and 100. The higher the value, the more intense the participants cravings are. Pre and post differences in craving will be assessed.
Effect of rTMS directed at left DLPFC on craving for methamphetamine as assessed by the Stimulant Craving Questionnaire (STCQ). | 6 weeks
  The Stimulant Craving Questionnaire-Brief (STCQ) is a 10-item self-report measure that assesses current craving for methamphetamine, using a seven-point scale, with answers ranging from 0 ("strongly disagree") to 6 ("strongly agree"). A composite score is generated for each participant by averaging the responses over all 10 questions. The scores can range from 0 to 6. The higher the composite score, the stronger the current craving. Pre and post differences in craving will be assessed.

SECONDARY OUTCOMES:
Effect of craving for methamphetamine on relapse status after rTMS directed at left DLPFC. | 5 months
  Relapse will be determined by self-report and/or positive urine drug screens.
Effect of cue type (methamphetamine versus neutral) on methamphetamine craving after rTMS treatment. | 6 weeks
  A composite craving score will be generated by adding each of the three craving measure scores (Severity of Dependence, Visual Analog Scale, and Stimulant Craving Questionnaire) for each participant who received real rTMS treatments. The composite score can range from 0 to 121, where 0 indicates no cravings for methamphetamine and 121 is the strongest possible cravings for methamphetamine. Pre and post differences in craving will be compared between participants who were exposed to methamphetamine cues before each session and those who were exposed to neutral cues.

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs Portland Health Care System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No